CLINICAL TRIAL: NCT00985699
Title: Pharmacogenomics of Oxidative Stress-Related Genes in Lymphoma
Brief Title: S8516-S8736-S9125-S9240 Research Study of Genes in Tissue Samples From Patients With B-cell Non-Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000643248; SWOG-S8516-S8736-S9125-S9240-S (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Lymphoma
Keywords: non-Hodgkin lymphoma; cutaneous B-cell non-Hodgkin lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone | interventions — Amplified Fragment Length Polymorphism Analysis; Pharmacogenomic Testing

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: pharmacogenomic studies

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at genes in tissue samples from patients with B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if toxicity following treatment for lymphoma varies according to genetic polymorphisms in oxidative stress-related genes (i.e., SOD2, CAT, GPX1, GSTM1, and GSTP1).
* To assess whether these genetic polymorphisms are associated with progression-free survival and/or overall survival in these patients treated for lymphoma.

OUTLINE: Previously collected samples are used for biomarker analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of aggressive B-cell non-Hodgkin lymphoma

  * Previously treated with curative intent using anthracycline-based therapies
* Previously collected paraffin-embedded diagnostic tissues from clinical trials that were collected as part of SWOG treatment protocols (S8516, S8736, S9125, S9240, and S9349) available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled on S8516 S8736 S9125 S9240 consenting to banking
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2009-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Association of polymorphisms in oxidative stress-related genes with overall survival and/or progression-free survival | retrospectively
Association of polymorphisms in these genes with rate of grade 4-5 hematologic toxicity | retrospectively

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M. Briehl, PhD, Study Chair — University of Arizona